CLINICAL TRIAL: NCT04748510
Title: A Prospective Randomised Control Trial Comparing the Effect of Functional Alignment With Mechanical Axis Alignment on Outcomes After Total Knee Arthroplasty.
Brief Title: Functionally Aligned vs Mechanical Axis Aligned Total Knee Arthroplasty
Acronym: FATKAvsMATKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perth Hip and Knee (Other)
Collaborators: St John of God Private Hospital Subiaco (Unknown)
Responsible Party: Principal Investigator, Gavin Clark, Principal investigator, Perth Hip and Knee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTRN12621000060842
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis; Osteo Arthritis Knee
Keywords: OA; Arthritis; Knee; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functionally aligned Total Knee Arthroplasty (Active Comparator): Knee arthroplasty performed using a functional alignment theory
  Interventions: Procedure: Functionally Aligned Total Knee Arthroplasty
- Mechanical axis aligned Total Knee Arthroplasty (Active Comparator): Knee arthroplasty performed using a mechanical alignment theory
  Interventions: Procedure: Mechanically Aligned Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Functionally Aligned Total Knee Arthroplasty — Femoral + tibial osteotomy planned for equal resection of femoral condyles to replicate patient anatomy. In coronal plane, distal femoral resection of 6.5mm subchondral bone from medial + lateral condyles, adjusted 1-3mm for compensation of wear. Proximal tibia, 7mm resection from subchondral bone from medial + lateral tibial plateau. Sagittal plane, resection angle determined intraoperatively to closely match native femoral flexion + tibial slope. Axial plane: posterior femoral resection 6.5mm from the subchondral bone of medial and lateral posterior condyles. Tibial rotation aligned to Akagi's line. Adjustments will be made to bony alignment to balance soft tissues within boundaries of 6° varus/3° valgus HKA alignment. Femoral component alignment limited to 6° valgus/3° varus in coronal plane. Tibial alignment limited 6° varus/3° valgus in coronal plane. Combined flexion of components limited to 10° flexion. Soft tissue release if balance within boundaries not achieved.
  Arms: Functionally aligned Total Knee Arthroplasty
Procedure: Mechanically Aligned Total Knee Arthroplasty — Tibial and femoral osteotomies in the coronal plane will be planned perpendicular to the tibial and femoral mechanical axes respectively to achieve neutral overall alignment. Soft tissue balance will be assessed and minor adjustments to bony alignment made to balance the knees with a maximal adjustment of two degrees valgus and two degrees varus of coronal alignment from neutral. Femoral rotation will be planned to surgical epicondylar axis and adjustments to rotation made to allow equal flexion and extension balance (to within 1mm). If balance can not be achieved within these boundaries then soft tissue release will be undertaken. In the sagittal plane, 0-3° degrees of posterior tibial slope and 0-5° of femoral component flexion will be used to optimise implant sizing whilst preventing notching. In the axial plane, the tibial component aligned to Akagi's line, which connects the medial border of the patellar tendon attachment to the middle of the posterior cruciate ligament.
  Arms: Mechanical axis aligned Total Knee Arthroplasty

SUMMARY:
The objective of this study is to compare clinical and radiological outcomes in robotic-arm assisted TKA using mechanical alignment (MA TKA) versus robotic-arm assisted TKA with functional alignment (FA TKA).

These outcomes will be used to determine if patient recovery is better with functionally aligned Mako robotic-assisted total knee arthroplasty (FA TKA) or mechanically aligned Mako robotic-assisted total knee arthroplasty (MA TKA).

DETAILED DESCRIPTION:
This project is being conducted by Perth Hip and Knee Clinic. The objective of this study is to compare clinical and radiological outcomes in robotic-arm assisted TKA using mechanical alignment (MA TKA) versus robotic-arm assisted TKA with functional alignment (FA TKA). Both FA TKA and MA TKA are performed through similar skin incisions, robotic-guidance, and use identical implants. In MA TKA, bone is prepared and implants positioned to ensure that the overall alignment of the leg is in neutral. In FA TKA, the bone is prepared and implants positioned to restore the natural alignment of the patient's leg. Both of these surgical techniques provide excellent outcomes in TKA but it is not known which of the two techniques is better for patient recovery. Mako robotic-assisted TKA is an established treatment for arthritis of the knee joint. The positions of the implants and overall alignment of the leg are important as they influence how quickly the implants wear out and need replacing. The aim of this study is to determine if patient recovery is better with functionally aligned Mako robotic-assisted total knee arthroplasty (FA TKA) or mechanically aligned Mako robotic-assisted total knee arthroplasty (MA TKA).

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptomatic knee osteoarthritis requiring primary TKA
* Patient and surgeon are in agreement that TKA is the most appropriate treatment
* Patient is fit for surgical intervention following review by surgeon
* Patient is between 45-75 years of age at time of surgery, computer literate, and able to complete patient-reported outcome measures independently.
* Patient must be capable of giving informed consent and agree to comply with the postoperative review program.
* Patient must be a permanent resident in an area accessible to the study site
* Patient must have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken
* Patient has tried non-pharmacologic therapies including: patient education, self-management programs, aerobic exercise, weight loss, physiotherapy and occupational therapy
* Patient has tried appropriate pharmacologic therapies including: regular paracetamol and NSAIDS if appropriate

Exclusion Criteria:

* Patient is not suitable for routine primary TKA. E.g., patient has ligament deficiency that requires a constrained prosthesis
* Interoperative requirement for a more constrained implant.
* Intraoperative requirement for the Posterior Cruciate Ligament to be released. These patients will be still included in the study, but analyzed with an intention-to-treat principle.
* Patient has bone loss that requires augmentation
* Patient requires revision surgery following previously failed correctional osteotomy or ipsilateral TKA (e.g., post-high tibial or distal femoral osteotomy)
* Patient requires a polyethylene inset of 13mm or greater.
* Patient is immobile or has another neurological condition affecting musculoskeletal function
* Patient is less than 44 years of age or greater than 76 years of age
* Patient is a compensable patient. I.e., Worker's compensation claim or motor vehicle accident.
* Patient is already enrolled in another concurrent clinical trial
* Patient is unable or unwilling to sign the informed consent form specific to this study
* Patient is unable to attend the follow-up program
* Patient is non-resident in local area or expected to leave the catchment area postoperatively
* Patients who lacks capacity to provide consent, or the ability to understand the study protocol due to a cognitive condition (e.g., Dementia)
* Patient is unable to communicate effectively in English.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Clark, Principal Investigator — Principal Investigator
Locations (2):
- Australia (2):
  - Perth Hip and Knee, Subiaco, Western Australia
  - St John of God Private Hopsital, Subiaco, Western Australia

IPD SHARING:
Plan to Share IPD: No
Not shared - for confidentiality of participants

REFERENCES:
- [Derived] Steer R, Tippett B, Khan RN, Collopy D, Clark G. A prospective randomised control trial comparing functional with mechanical axis alignment in total knee arthroplasty: study protocol for an investigator initiated trial. Trials. 2021 Aug 9;22(1):523. doi: 10.1186/s13063-021-05433-z. PMID 34372888

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Functionally Aligned Total Knee Arthroplasty | Mechanical Axis Aligned Total Knee Arthroplasty
Started | 50 | 50
Completed | 48 | 44
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Population: 100 cases were randomised. 1 MA case was then removed from cohort analysis due to protocol changes in alignment technique during surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Functionally Aligned Total Knee Arthroplasty | Mechanical Axis Aligned Total Knee Arthroplasty | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (6.2) | 65.4 (7.3) | 65.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 52
  Male | 22 | 25 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (6.4) | 31.0 (5.2) | 31.2 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Forgotten Joint Score After 2 Years From Baseline
Description: Difference in relative change in Forgotten Joint Score (2 years post-operatively compared to preoperatively) between FA and MA patients. Scale 0-100 with higher scores being a better outcome
Time Frame: Preoperatively and 2 years postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functionally Aligned Total Knee Arthroplasty | Mechanical Axis Aligned Total Knee Arthroplasty
Number analyzed (Participants) | 48 | 44
score on a scale | 50.1 (28.3) | 46.4 (32.4)

2. Primary Outcome: Change in Oxford Knee Score After 2 Years From Baseline
Description: Difference in relative change in Oxford Knee Score (2 years post-operatively compared to preoperatively) between FA and MA patients. Scale 0-48 with higher scores being a better outcome.
Time Frame: Preoperatively and 2 years postoperatively
Population: 11 patients did not provide responses for this outcome measure, resulting in missing scores. Some of these participants did complete other study questionnaires but were lost to follow-up for this specific assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functionally Aligned Total Knee Arthroplasty | Mechanical Axis Aligned Total Knee Arthroplasty
Number analyzed (Participants) | 45 | 43
score on a scale | 17.0 (7.5) | 17.2 (8.6)

3. Primary Outcome: Change in Range of Motion After 2 Years From Baseline
Description: Difference in relative change in range of motion via goniometry (2 years post-operatively compared to preoperatively) between FA and MA patients.
Time Frame: Preoperatively and 2 years postoperatively
Population: 18 participants were lost to in-person clinical follow-up, resulting in missing range-of-motion scores. Reasons for loss to follow-up included cancer diagnosis, relocation outside the Perth metropolitan area, appointment cancellations or refusals, and inability to contact the participants. However, some of these individuals completed the study questionnaires and were lost to follow-up only for the range-of-motion assessment.
Measure: Mean (Standard Deviation); unit: deg
Arm/Group | Functionally Aligned Total Knee Arthroplasty | Mechanical Axis Aligned Total Knee Arthroplasty
Number analyzed (Participants) | 40 | 41
deg | 2.8 (9.9) | 2.8 (9.3)

4. Secondary Outcome: Determine Lower Limb Alignment Achieved With Both Alignment Techniques
Description: Lower limb alignment as assessed using standing long leg x-rays performed postoperatively at 3 months. Measurements of the hip-knee-angle (HKA), medial proximal tibial angle (MPTA) and lateral distal femoral angle (LDFA). Also evidence of imbalance with implant lift off will be measured.
Time Frame: 3 Months post-operatively
Reporting Status: Not Posted

5. Secondary Outcome: Difference in Analgesia Requirements Between Patients in Alignment Groups
Description: Determine if there are any differences in analgesic requirements based on alignment method used.
  Inpatient medical records will be utilised to obtain analgesia requirements as inpatient Questionnaires will be used to obtain analgesia usage at remaining timepoints. Analgesia usage will be converted to morphine equivalent dosages for comparison
Time Frame: 6 weeks, 3 months, 1 year, 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Difference in Sagittal Stability of the Knee Post Replacement
Description: Determine whether alignment method utilized has an effect on the sagittal stability of the knee post replacement, as measure with an arthrometer "Lachmeter"
Time Frame: Preop, and post-operatively at 3 months, 1 year and 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Difference in Functional Outcomes (Measured as Maximal Voluntary Contraction) of Knee Flexion and Extension Between Alignment Groups
Description: Determine whether alignment method utilized has an effect on functional outcomes.
  Measured as Maximal voluntary isometric knee flexion and extension forces as measured via hand-held dynamometry.
Time Frame: Preop, 3 months, 1 Year and 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Intra-operative Balance Achieved With Different Alignment Techniques.
Description: Surgeon blinded measurement of intraoperative balance achieved with Verasense sensor (smaller cohort) Secondary outcome [6] To determine if there is a difference in knee kinematics between the two techniques. Measurement of knee kinematics with Verasense sensor to assess presence or absence of medial pivot (smaller cohort)
Time Frame: Intraoperatively
Reporting Status: Not Posted

9. Secondary Outcome: Difference in Clinical Outcomes as Measured in Knee Injury and Osteoarthritis Outcome Score for Joint Replacement Score (KoosJR)
Description: Difference in operated knee outcome on Koos JR scale between FA and MA patients. Scale 0-100 where higher scores mean better outcome.
Time Frame: Measured Pre-operatively and at 3 month, 1 year and 2 years post operatively.
Reporting Status: Not Posted

10. Secondary Outcome: Difference in Clinical Outcomes as Measured in European Quality of Life Questionnaire With 5 Dimensions for Adults (EQ-5D-5L).
Description: Difference in overall by Visual Analogue Scale for overall health (VAS). Scale: Five dimensions combined into a 5-digit number lower numbers represent better outcomes. Addition of overall health VAS Scale 0-100 with higher score being better outcome.
Time Frame: Measured Pre-operatively and at 3 month, 1 year and 2 years post operatively.
Reporting Status: Not Posted

11. Secondary Outcome: Difference in Operated Knee Pain as Measured by Visual Analogue Scale for Pain (VAS)
Description: Difference in operated knee pain as measured by Visual Analogue Scale for pain (VAS). Scale 0-100 with higher scores meaning worse outcome.
Time Frame: Measured Pre-operatively and at 3 month, 1 year and 2 years post operatively.
Reporting Status: Not Posted

12. Secondary Outcome: Difference in Clinical Outcomes as Measured by Kujala Score- a Measure of Anterior Knee Pain and Best Clinical Score for Patellofemoral Function
Description: Difference in clinical outcomes as measured by Kujala score between FA and MA patients. Scale 0-100, with higher scores indicating better outcome.
Time Frame: Measured Pre-operatively and at 3 month, 1 year and 2 years post operatively.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each participant from the time of enrolment (baseline) through to their final study visit (2 years post-operative).
Description: Both methods of knee alignment are already being performed as standard of care for both surgeons. There are no additional risks to the patient stemming from either trial intervention, apart from routine risk of surgery.
Arm/Group | Functionally Aligned Total Knee Arthroplasty | Mechanical Axis Aligned Total Knee Arthroplasty
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functionally Aligned Total Knee Arthroplasty (N=50) | Mechanical Axis Aligned Total Knee Arthroplasty (N=49)
MUA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Paroxsymal SVT post operative (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT04748510/Prot_SAP_ICF_000.pdf